## **ConnectED ICF**

Study Title: Connect\_ED

| Institution/Site: | University of Kentucky |
|----------------------------------|------------------------|
| Document (Approval/Update) Date: | 03/04/18 |
| NCT Number: | NCT02786472 |
| IRB Number | 15-0856-P1H |
| Coversheet created: | 02/19/20 |

## **Global Link**

Thank you for your interest in Connect ED!

Connect\_ED is a CDC (Centers for Disease Control and Prevention) funded study looking at the effectiveness of different training programs to improve new UK students' life skills. New UK undergraduate students age 17-24 are eligible for this research study. Consenting students receive training emphasizing strategies to prevent or reduce the risk of interpersonal violence or substance abuse for students enrolled at UK.

If you agree to study participation you will be one of the first students to participate in this study and training program, and your participation in Connect\_ED would be for this academic year.

Study participation includes

- Completing a 90 minute educational training,
- Completing 3 brief surveys (5-10 minutes), and
- Responding to smartphone surveys via MyUK app or text message/push notification

You have a choice to participate in this study. If you agree to participate and complete this contact information form, you will be randomly assigned to participate in a training at either the Fall or Spring semester, which will take 90 minutes to complete. All trainings will take place on UK's campus and times and locations of training will be sent to you via email or text. You will receive a \$40 gift card for completing the first brief survey and the assigned training. In the Fall and Spring semesters, you will receive an invitation to complete two short, follow-up surveys (takes about 5-10 minutes). You will be offered \$5 to your PLUS Account for completion of each of these two short surveys. These surveys will ask about experiences that you may have encountered while at college. Throughout the academic year, you will also receive push notifications to answer questions on your smartphone via text or MyUK App. If you complete all smartphone surveys you will additionally receive \$10 dollars via your PLUS Account. Completing all follow up and smartphone surveys will result in a total of \$20 via your PLUS account.

Although we have tried to minimize this, some questions may make you upset or feel uncomfortable and you may choose not to answer them. If some questions do upset you, we will provide information on campus and community resources that may help you with these feelings.

All answers that you give will be kept private. This is because this study has been given a Certificate of Confidentiality. This means anything you tell us will not have to be given out to anyone, even if a court orders us to do so, unless you say it's okay. But under the law, we must report to the proper authorities suspected cases of child abuse or if you tell us you are planning to cause serious harm to yourself or others. When we write about the results of the study, you will not be identified and your responses will be confidential. Please be aware, while we make every effort to safeguard your data once received on our servers via REDCap, given the nature of online surveys, as with anything involving the Internet, we can never guarantee the confidentiality of the data while still en route to us. Because of recent changes in computer technology your answers may be linked with other data. Examples of types of other data include student records and previous surveys conducted by the university. Any linked data would not name you or provide any identifying information like your address, phone or social security number.

If you have questions about the study, please feel free to ask our research coordinator Kelsey Rutheford at Connect\_ED@uky.edu or our principal investigators Heather Bush at heather.bush@uky.edu or Ann L. Coker at ann.coker@uky.edu. If you have complaints, suggestions, or questions about your rights as a research volunteer, contact the staff in the University Office of Research Integrity at (859) 257-9428 or toll-free at 1-866-400-9428.

Thank you in advance for your help with this important project.

The first electronic survey takes about 5-10 minutes to complete. You need to complete this survey to be eligible for training. You may prefer to complete this survey in a private setting. This survey link will be sent to you later.

| Thanks,<br>Connect_ED<br>Email: Connect_ED@uky.edu<br>Please save or print a copy of this letter for your records. |
|---|
| Do wish to participate in this study? |
| Yes, I wish to participate. |

**REDCap** 

03/04/2018 9:07pm

No, I do not wish to participate.